# 知情同意书

研究名称: 自体瘢痕真皮支架的组织工程皮肤移植修复增生性瘢痕的多中心随机对照 临床试验

| 项目负责人: | 电话: | |
|----------------|-------------------|-------|
| 您将被邀请参加一项临床研究。 | 本知情同意书提供给您一些信息以帮助 | 助您决定是 |

您将被邀请参加一项临床研究。本知情同意书提供给您一些信息以帮助您决定是 否参加此项临床研究。请您花时间仔细阅读,如有任何疑问请向研究医生或工作人员 提出。

## 关于此项研究:

## 1. 研究目的:

这是一项评估自体表皮基底细胞结合自体真皮支架复合移植修复增生性瘢痕的多中心随机对照临床试验的安全性和有效性的研究。旨在提高增生性瘢痕植皮的成活率,同时改善植皮愈后,进一步改善患者生活质量。

增生性瘢痕的修复一直以来是临床中的难题,目前皮片移植修复创面的金标准,但是,取皮区遗留瘢痕。如果采用复合皮移植,植皮成活率偏低,皮源不足。因此,我们结合临床实践经验,以及前期的临床研究(已发表在国际著名杂志 Brit J Surg上),应用自体表皮基底细胞复合自体真皮支架和自体皮片修复增生性瘢痕,有望解决增生性瘢痕修复的难题。此项研究已获得中山大学附属第一医院医学伦理委员会的批准。部分相关经费将由中山大学临床医学研究 5010 计划提供。

#### 2. 研究过程

可能存在某些原因导致您不能参加此项研究。其中部分原因包括:

- 己存在的疾病会影响到植皮成活(恶性肿瘤、自身免疫病)
- 需使用大剂量糖皮质激素(即每日接受≥ 40 mg 泼尼松或泼尼松等量,为期≥ 2 周)影响创面愈合
- 有严重未控制的疾病或全身急性感染者及合并其他严重心、肺、脑病等严重脏器 疾病者
- 不能配合临床试验人员完成试验者
- 正在怀孕或哺乳,或计划在本研究期间怀孕或哺乳
- 之前参与过本研究。

研究医生将对这些原因以及其它任何导致您不得入选研究的原因进行讨论。将有大约 226 人参加这项研究。您参加这项研究的持续时间约为 12 个月。

参加此项研究后,您需要遵循以下要求:

- 研究期间需要到医院随访 3 次。最后一次随访是在植皮手术后 12 个月,进行安全性随访和有效性评估。
- 在接受手术前,将会常规抽血进行相关实验室安全性检查,待检查完善后,再行 瘢痕切除植皮手术。
- 育龄期妇女及其伴侣必须使用充分的避孕方法或同意停止性活动。这必须从第一次研究访视持续到手术后 1 个月。充分的避孕方法包括口服避孕药、子宫内避孕器(IUD)、带有杀精子剂的避孕隔膜、避孕海绵、避孕套和输精管切除术。
- 在接受植皮手术时,将随机分配(分配到各组概率为50%)到试验组(自体表皮基底细胞复合自体真皮支架和自体皮片移植)或对照组(传统自体皮片移植),术后1周、2周分别进行访视。
- 在手术后,需要观察植皮区情况,如果有任何不适,请告诉您的研究医生。 在研究期间的随访中,研究医生或工作人员可能会进行以下任何一项或所有步骤:
- 在您开始接受任何研究的操作之前,将会通过签署本知情同意书询问您是否同意 参与本研究。
- 研究医生将会决定您是否适合入选本研究并接受手术。
- 回顾您的病史。
- 评估和并记录您创面的情况。
- 审查并记录您正在使用的药物。
- 询问上次访视以来是否出现任何创伤或疾病
- 评估和记录一般生命体征和术区情况以上某些检查是用于评价手术的有效性,另外一些是用于监测您的健康状况。

#### 3. 可能的风险

在进行某些检查时您可能感觉不适,也可能有一定风险,例如:

- 一般的手术风险包括麻醉意外、出血、感染等。
- 植皮失活。

以上风险发生概率极低,通过有效的预防措施和全面的术前筛查准备,将可有效避免发生。据前期研究以及目前文献资料显示,自体皮片移植是增生性瘢痕修复的一线治疗方法,如出现植皮失活,将择期行二期手术修复。

#### 4. 可能的不良反应

在进行治疗的过程中,有可能局部或全身出现皮疹、搔痒或其它过敏现象,或局部出现红、肿、热、痛的感染症状,或植皮区出现皮片溶解坏死。

针对以上可能出现的不良反应,我们有丰富的临床经验和相应的处理对策,可最 大限度减轻伤害。如果发生严重急性过敏反应,可能需要使用皮下肾上腺素和其他急 救措施。如果您有关于不良反应的任何问题,请告知您的研究医师。

#### 5. 受试者收益

本次临床观察试验方案要求的部分相关临床检验检查项目、部分随访交通费将由我方免费提供。对遵循临床试验方案的患者所发生与试验有关的损害承担相应的治疗费用及相应的经济补偿。

本次临床观察试验将免费提供自体细胞提取相关耗材给实验组受试者。随访时可能产生一些额外费用比如交通费、停车费等,这些合理的和本研究相关的费用,如果您提供正式发票给研究医师,将得到相应的交通费用补贴(12个月随访完成后受试者最高可获得人民币 500 元的交通补偿)。对遵循临床试验方案的患者所发生与试验有关的损害承担相应的治疗费用及相应的经济补偿。

参加此项研究您无任何报酬。

#### 6. 研究记录的保密

如果您决定参加本项研究,研究医生及其他研究人员将使用您的医疗信息进行研究。这些信息可能包括您的姓名、地址、电话号码、病史及在您研究随访时得到的信息。这些医疗信息可能来源于您的家庭医生或其他医疗保健工作者。

你提供的信息将在以下情况下被用到:

- 研究过程中涉及到的行政管理需要
- 规章条例需要,包括为了顺应 SFDA 的相关条例
- 透露给那些与你的治疗相关的人,包括你的主管医生和监护人。当有需要时,这些信息可能会透露给别的医生,或以医学研究及报告的方式透露给相关专业人士。如公开发表试验结果,也会对受试者的身份保密。

#### 7. 受试者的权利

受试者参加此试验是自愿的,受试者可以拒绝参加或在试验的任何阶段,随时退出试验而不会遭到歧视或报复,其医疗待遇与权益不受影响。

如果您不想参加本项研究,还有如下选择:

脱细胞异体真皮复合皮移植,皮瓣移植等。

研究医生会与您讨论这些选择。您不是必须参与本项研究治疗您的溃疡。

### 8. 受试者声明

在签署了知情同意书后, 我将同意:

- 我已经阅读了本知情同意书。
- 我有机会提问而且所有问题均已得到解答。
- 我理解参加本项研究是自愿的。
- 根据本同意书上所描述,同意使用及分享我的医疗信息,但不使用受试者的名字。
- 我可以选择不参加本项研究,或者在任何时候通知研究医生后退出。我将不会因此 受罚或丧失任何应有的利益。同时这并不会影响常规治疗。
- 如果我需要其它治疗,或者我没有遵守研究计划,或者发生了与研究相关的损伤或者有任何其它原因,可以不得到我的同意而被退出本项研究。
- 如果因任何原因我退出本项研究,研究医生可能要求为我做一些最后的检查。
- 谈话医师已将相关内容向我详细介绍,我对本次谈话内容充分知情理解,并且确 认对手术相关情况及手术可能发生的意外风险或并发症表示知情和理解,并对医院和 经治医师的工作表示信任。我愿意承担手术风险,同意进行手术。

| 患者或委托人签名: | 日期: | _ |
|-----------|-----|---|
| 医师签名: | 日期: | |